CLINICAL TRIAL: NCT06841523
Title: Intelligent Pressure and Temperature Control Ureteral Soft Scope System for the Treatment of Upper Ureteral Stones Complicated With Infection in the Kidney and Upper Ureter: a Multicenter Randomized Controlled Clinical Study
Brief Title: An Intelligent Pressure and Temperature Control Ureteral Soft Scope System for Treating Stones With Infection.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xu Kewei, Principal Investigator, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-1120-02
Record Dates: First submitted 2025-02-09; First posted 2025-02-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ureterolithiasis; Renal Calculi
Keywords: Ureteral Stone; renal stone; Ureteroscopy; Upper urinary tract stones with concurrent infection
MeSH Terms: conditions — Ureterolithiasis; Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Arm 1: Intelligent Pressure and Temperature-Controlled Ureteroscope System Arm 2: Conventional Ureteroscope
Who Masked: Participant
Masking Description: Prior to the surgery, it is necessary to select the surgical technique and follow the trial protocol by opening an envelope in the specified sequence. This trial protocol follows a "single blind" format, meaning that the researcher is aware of the surgical method while the subject remains unaware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intelligent Pressure and Temperature-Controlled Ureteroscope System (Active Comparator): Participants in this arm will undergo surgery using the Intelligent Pressure and Temperature-Controlled Ureteroscope System, which monitors and adjusts intrarenal pressure and temperature in real-time to ensure safe and effective lithotripsy.
  Interventions: Device: Intelligent Pressure and Temperature-Controlled Ureteroscope System
- Conventional Ureteroscope (Active Comparator): Participants assigned to this arm will undergo surgery with a conventional ureteroscope. The procedure involves standard ureteroscopic lithotripsy without real-time pressure or temperature monitoring.
  Interventions: Device: Conventional Ureteroscope

INTERVENTIONS:
Device: Intelligent Pressure and Temperature-Controlled Ureteroscope System — RIRS procedure for upper ureteral or renal stone lithotripsy with Intelligent Pressure and Temperature-Controlled Ureteroscope System
  Arms: Intelligent Pressure and Temperature-Controlled Ureteroscope System
Device: Conventional Ureteroscope — RIRS procedure for upper ureteral or renal stone lithotripsy with conventional ureteroscope
  Arms: Conventional Ureteroscope

SUMMARY:
The goal of this clinical trial is to determine the efficacy and safety of a novel intelligent pressure and temperature-controlled ureteroscope system for treating renal and upper ureteral stones with concurrent infection. It will also assess its ability to reduce postoperative complications and improve stone clearance rates. The main questions it aims to answer are:

Does the intelligent system lower the complication rate and enhance stone clearance compared to standard ureteroscopy? What safety issues or medical problems do participants experience when using the intelligent system? Researchers will compare the intelligent pressure and temperature-controlled ureteroscope system to a standard ureteroscope to evaluate its effectiveness in treating renal and upper ureteral stones.

Participants will:

Undergo surgery using either the intelligent system or a standard ureteroscope Be monitored for postoperative complications, stone clearance, and other relevant outcomes Participate in follow-up visits to assess recovery and treatment efficacy

DETAILED DESCRIPTION:
This study protocol describes a multi-center, prospective, randomized controlled trial with a non-inferiority design, aiming to assess the efficacy and safety of an intelligent pressure and temperature-controlled ureteroscope system for treating renal and upper ureteral stones with concurrent infection. A total of 288 patients will be randomized into two groups (1:1 ratio), with the intervention group receiving the intelligent system and the control group undergoing standard ureteroscopy. The primary endpoints are the complication rate and stone clearance rate at 1 month postoperatively, while secondary endpoints include short-term stone clearance, intraoperative and postoperative complications, infection markers, surgical time, and intraoperative pressure and temperature monitoring. The study will adhere to rigorous ethical standards and statistical analysis plans to provide robust evidence for the clinical application of this novel device.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ Age ≤ 75 years old, regardless of gender, able to tolerate surgery;
2. ASA I-III;
3. Patients who have been confirmed by bilateral renal/urinary tract CT to have upper ureteral or renal stones, single or multiple, with a cumulative maximum diameter of 10mm < cumulative maximum diameter ≤ 20mm, and are planning to undergo ureteroscopic lithotripsy for stone removal;
4. Confirmed urinary tract infection, indicated by positive urine leukocytes and nitrite, or positive urine culture, with appropriate antibiotic treatment administered preoperatively;
5. Those who voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. Uncontrollable systemic hemorrhagic disease;
2. Severe spinal deformities, severe hip joint deformities, and difficulty in lithotomy position;
3. Uncontrolled acute urinary tract infections;
4. Any intracavitary surgery caused by anatomical factors of the urinary system cannot be performed;
5. Pregnant, planned pregnancy within 3 months, and lactating female patients;
6. The patients determined by the investigator to be unsuitable for this study include (but are not limited to): known to have human immunodeficiency virus (HIV) or AIDS; Suffering from mental illness; Infectious diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication Rate | Assessed at 48 hours and 1 month postoperatively.
  This composite outcome measure includes the incidence of the following complications:
  1. Fever: Defined as body temperature ≥38℃.
  2. Urinary Sepsis: An increase in the Sequential Organ Failure Assessment (SOFA) score by ≥2 points postoperatively.
  3. Septic Shock: Requires vasopressors to maintain mean arterial pressure ≥65 mmHg after adequate fluid resuscitation, with blood lactate concentration >2 mmol/L
  4. Pain: Assessed using the Numeric Rating Scale (NRS) within 48 hours postoperatively, recording the need for Nonsteroidal Anti-inflammatory Drugs (NSAIDs) or other analgesic treatment.
  5. Renal subcapsular or perirenal hematomaL: Diagnosed by Computed Tomography (CT) or other imaging within 30 days postoperatively.
  The composite postoperative complication rate will be calculated as the number of patients with at least one complication divided by the total number of patients in the study, multiplied by 100 to obtain a percentage.
Stone Free Rate | Assessed at 1 month postoperatively.
  This is defined as the proportion of patients with no residual stones or residual stones ≤2mm in diameter and asymptomatic, as confirmed by renal CT at 1 month postoperatively.

SECONDARY OUTCOMES:
Stone Clearance Rate at 48 hours postoperatively | Assessed at 48 hours postoperatively.
  The proportion of patients with no residual stones or residual stones ≤2mm in diameter and asymptomatic, as confirmed by renal CT at 48 hours postoperatively.
Intraoperative Complications Rate | Assessed at 2 hours after the surgical procedure.
  The incidence of intraoperative complications, including ureteral or renal pelvis perforation, ureteral mucosal stripping, ureteral rupture, the need for conversion to other treatments, and failure of ureteral access sheath placement.
Concentration of postoperative infection markers | Assessed at 48 hours postoperatively during hospitalization.
  Changes in the concentration of postoperative infection markers Procalcitonin (PCT) and C-reactive protein (CRP), hemoglobin (Hb), serum creatinine (Scr), and blood urea nitrogen (BUN).
Intraoperative Pressure | Assessed 2 hours after the surgical procedure.
  The intraoperative pressure values recorded during the procedure measured by the intelligent pressure and temperature control ureteral soft scope system.
Intraoperative Temperature | Assessed at 2 hours after the surgical procedure.
  The intraoperative temperature values recorded during the procedure.
Postoperative Hospital Stay | Assessed at 24 hours after patients leaving the hospital
  The length of hospital stay following the surgical procedure.
Surgical and Lithotripsy Time | Assessed at 24 hours postoperatively.
  The duration of the surgical procedure and the time required for lithotripsy.

CONTACTS AND LOCATIONS:
Overall Officials: Kewei Xu, MD, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No